CLINICAL TRIAL: NCT04527146
Title: GEnetic Counseling Through VIRTUAL Visits in Parkinson's Disease
Acronym: GET-VIRTUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Thomas Tropea, DO, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 843748; PCPM (Other: Penn Center for Precision Medicine)
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized into one of 4 groups based on pre- and post-genetic test counseling: (1)IMAGINE-PD/Virtual, (2)IMAGINE-PD/Telephone, (3)Virtual/Virtual, and (4)Virtual/Telephone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IMAGINE-PD/Virtual (Experimental): Pre-test genetic counseling through the Interactive Multimedia Approach to Genetic counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) website. Genetic results disclosure via virtual visit with a genetic counselor.
  Interventions: Other: IMAGINE-PD; Other: Virtual genetic counseling
- IMAGINE-PD/Telephone (Experimental): Pre-test genetic counseling through the Interactive Multimedia Approach to Genetic counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) website. Genetic results disclosure via telephone with a genetic counselor.
  Interventions: Other: IMAGINE-PD; Other: Telephone genetic counseling
- Virtual/Telephone (Experimental): Pre-test genetic counseling virtual visit with a genetic counselor. Genetic results disclosure via telephone with a genetic counselor.
  Interventions: Other: Virtual genetic counseling; Other: Telephone genetic counseling
- Virtual/Virtual (Active Comparator): Pre-test genetic counseling and genetic results disclosure via virtual visit with a genetic counselor.
  Interventions: Other: Virtual genetic counseling

INTERVENTIONS:
Other: IMAGINE-PD — The Interactive, Multimedia Approach to Genetic Counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) is a novel, interactive, web-based, audiovisual, self-guided, genetic counseling tool in the development phase. Essential genetic counseling themes, outlined by a senior certified clinical genetics counselor in accordance with national guidelines, are presented in a web-based format, utilizing videos, text, pictures, and audio. Participants can interact with IMAGINE-PD at their own pace, with the ability to move backward and forward, repeat sections, and have the ability to submit questions to the genetic counselor via e-mail.
  Arms: IMAGINE-PD/Telephone; IMAGINE-PD/Virtual
Other: Virtual genetic counseling — The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans) within the Penn Chart/Epic electronic medical record dashboard.
  Arms: IMAGINE-PD/Virtual; Virtual/Telephone; Virtual/Virtual
Other: Telephone genetic counseling — The telephone counseling will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors.
  Arms: IMAGINE-PD/Telephone; Virtual/Telephone

SUMMARY:
The research study is being conducted to compare methods of virtual genetic counseling for people with Parkinson's disease.

DETAILED DESCRIPTION:
This research will evaluate different virtual methods of pre-test genetic counseling and post-test genetic results disclosure in people with Parkinson's disease. Participants will be randomized to receive different methods of genetic counseling using web-based, telephone, or telehealth methods. In both pre- and post-test counseling phases, remote genetic counseling methods will be compared to demonstrate equivalence. The primary outcomes will be equivalence on genetics knowledge and outcomes scales, and the revised impact of events scale. The purpose is to develop effective and scalable approaches to genetic counseling. This work is crucial for patient safety and will improve access to care through novel genetic counseling approaches.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to have clinical confirmation genetic testing, and comply with all study procedures and availability for the duration of the study
* Male or female, over the age of 21.
* English Speaking

Exclusion Criteria:

* Prior genetic counseling and/or clinical testing specifically for Parkinson's disease
* Montreal Cognitive Assessment (MoCA) < 21, or a prior diagnosis of dementia during the screening phase

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Tropea, DO, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Parkinsons Disease and Movement Disorders Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All data and isolated DNA samples will be stored for future research purposes for an indefinite amount of time. Individual participant data (IPD) may be shared with other research, academic, and medical institutions, other researchers, drug and device companies, biotechnology companies and others. In the event of such a collaboration, no personally identifying information will be shared. Potential collaborators may apply with a description of the proposed project. This application is then evaluated by a Biospecimen Review Access Committee (BRAC). Only projects deemed to have scientific or clinical merit will be considered eligible to receive samples or information, from which personally identifying information will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request by collaborators and upon publication of scientific manuscripts.
Access Criteria: Approval by the BRAC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants from UPenn's Parkinson's Disease and Movement Disorders Center's Molecular Integration in Neurological Diagnosis (MIND) Initiative who were 21 years old or older, willing to complete confirmatory genetic testing, willing to learn their genetic test results, and had access to a telephone, computer, and videoconferencing device. Key exclusion criteria were prior genetic counseling for PD, prior diagnosis of dementia, or scored <21 on the Montreal Cognitive Assessment (MoCA).
Pre-assignment Details: A factorial design schema was used for group randomization based on pre-test education or counseling (i.e., IMAGINE-PD or Virtual) and post-test counseling (i.e. Telephone or Virtual) modalities. All randomized participants were included in an intention-to-treat (ITT) analysis. A per protocol (PP) analysis defined a subset of participants with data for all 3 primary outcome variables (i.e., completed visit 3 for genetic counseling satisfaction, genetics knowledge, and test-related distress).
Groups:
- IMAGINE-PD/Virtual: Pre-test genetic education through the Interactive Multimedia Approach to Genetic counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) website. Genetic results disclosure via virtual visit with a genetic counselor.
  IMAGINE-PD: The Interactive, Multimedia Approach to Genetic Counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) is a novel, interactive, web-based, audiovisual, self-guided, genetic counseling tool in the development phase. Essential genetic counseling themes, outlined by a senior certified clinical genetics counselor in accordance with national guidelines, are presented in a web-based format, utilizing videos, text, pictures, and audio. Participants can interact with IMAGINE-PD at their own pace, with the ability to move backward and forward, repeat sections, and have the ability to submit questions to the genetic counselor via e-mail.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans or Zoom).
- Virtual/Telephone: Pre-test genetic counseling virtual visit with a genetic counselor. Genetic results disclosure via telephone with a genetic counselor.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans) within the PennChart/EPIC electronic medical record dashboard.
  Telephone genetic counseling: The telephone counseling will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors.
- Virtual/Virtual: Pre-test genetic counseling and genetic results disclosure via virtual visit with a genetic counselor.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors, in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans or Zoom).
Period: Overall Study
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Started (Randomized (ITT)) | 94 | 91 | 92 | 93
Completed (Completed all primary outcomes) | 61 | 63 | 65 | 60
Not Completed | 33 | 28 | 27 | 33
Not completed — Withdrawal by Subject | 12 | 15 | 7 | 16
Not completed — Lost to Follow-up | 13 | 9 | 16 | 13
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Ineligible after randomization | 2 | 0 | 2 | 2
Not completed — Moved to a different group | 6 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- IMAGINE-PD/Virtual: Pre-test genetic counseling through the Interactive Multimedia Approach to Genetic counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) website. Genetic results disclosure via virtual visit with a genetic counselor.
  IMAGINE-PD: The Interactive, Multimedia Approach to Genetic Counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) is a novel, interactive, web-based, audiovisual, self-guided, genetic counseling tool in the development phase. Essential genetic counseling themes, outlined by a senior certified clinical genetics counselor in accordance with national guidelines, are presented in a web-based format, utilizing videos, text, pictures, and audio. Participants can interact with IMAGINE-PD at their own pace, with the ability to move backward and forward, repeat sections, and have the ability to submit questions to the genetic counselor via e-mail.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans or Zoom).
- Virtual/Telephone: Pre-test genetic counseling virtual visit with a genetic counselor. Genetic results disclosure via telephone with a genetic counselor.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans or Zoom).
  Telephone genetic counseling: The telephone counseling will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors.
- Virtual/Virtual: Pre-test genetic counseling and genetic results disclosure via virtual visit with a genetic counselor.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans or Zoom).
- Total: Total of all reporting groups
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual | Total
Number analyzed (Participants) | 94 | 91 | 92 | 93 | 370
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [62 to 75] | 68 [64 to 73] | 68 [64 to 73] | 70 [60 to 74] | 69 [63 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 32 | 29 | 26 | 131
  Male | 50 | 59 | 63 | 67 | 239
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 1 | 6
  White | 88 | 88 | 88 | 85 | 349
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 94 | 91 | 92 | 93 | 370
PD family history [Count of Participants; unit: Participants]
  Yes | 33 | 42 | 38 | 37 | 150
  No/Unk/Missing | 61 | 49 | 54 | 56 | 220
Genetic Screening Result [Count of Participants; unit: Participants]
  Negative | 80 | 70 | 71 | 82 | 303
  Positive | 14 | 21 | 21 | 11 | 67
Education [Count of Participants; unit: Participants]
  < HS | 1 | 0 | 0 | 2 | 3
  HS | 2 | 7 | 4 | 5 | 18
  Associate | 12 | 14 | 17 | 15 | 58
  Bachelor | 34 | 34 | 30 | 28 | 126
  Graduate | 44 | 34 | 39 | 39 | 156
  Missing | 1 | 2 | 2 | 4 | 9
Disease Duration [Median (Inter-Quartile Range); unit: years] | 6 [4 to 11] | 6 [3 to 9] | 7 [1 to 12] | 7 [4 to 11] | 7 [3 to 11]
Baseline Genetics Knowledge (GKS) total [Median (Inter-Quartile Range); unit: units on a scale] — 20 question, true/false questionnaire, self-administered. Novel instrument adapted from questionnaires previously administered in PD research studies. Topics include general and PD-specific genetics knowledge, genetic testing attitudes and beliefs, interest in genetic testing and counseling.
  units on a scale | 16 [14 to 18] | 17 [15 to 19] | 17 [15 to 18] | 16 [15 to 18] | 17 [15 to 18]
Baseline Montreal Cognitive Assessment (MoCA) total [Median (Inter-Quartile Range); unit: units on a scale] — The Montreal Cognitive Assessment is a 30-point, validated cognitive screening tool. Test is administered by coordinator. Scores are added for a total (score range 0-30). Higher scores associate with better cognitive performance.
  units on a scale | 27 [25 to 28] | 27 [26 to 28] | 27 [25 to 28] | 26 [24 to 28] | 27 [25 to 28]
Baseline Geriatric Depression Scale (GDS) total [Median (Inter-Quartile Range); unit: units on a scale] — The Geriatric Depression Scale (short version) is a 15-item, "Yes/No", validated, self-report measure of depression in older adults.
  units on a scale | 3 [1 to 6] | 2 [1 to 5] | 2 [1 to 5] | 3 [1 to 5] | 3 [1 to 5]
Baseline State-Trait Anxiety Scale (STAI)-state [Median (Inter-Quartile Range); unit: units on a scale] — The State-Trait Anxiety Inventory is a 40 item, 4-point, well-validated self-report scale measuring aspects of both state- and trait-anxiety.
  units on a scale | 36 [30 to 43] | 37 [29 to 46] | 36 [30 to 46] | 36 [26 to 44] | 36 [29 to 45]
Baseline State Trait Anxiety Scale (STAI)-trait [Median (Inter-Quartile Range); unit: units on a scale] — The State-Trait Anxiety Inventory is a 40 item, 4-point, well-validated self-report scale measuring aspects of both state- and trait-anxiety.
  units on a scale | 35 [29 to 42] | 34 [28 to 42] | 34 [26 to 45] | 35 [29 to 43] | 34 [28 to 43]
Baseline Parkinsons Disease Questionnaire-39 (PDQ-39) item summary index (PDQ-39) [Median (Inter-Quartile Range); unit: units on a scale] — The PDQ-39 is a disease-specific health status measure that assess multiple dimensions of daily living. It is a validated, self-report measure for people with PD.
  units on a scale | 20 [11 to 32] | 18 [11 to 29] | 18 [7 to 32] | 19 [12 to 28] | 19 [10 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Genetics Knowledge
Description: Genetics Knowledge Scale (20-question true/false questionnaire, score range 0-20, higher scores mean greater knowledge)
Time Frame: 4 weeks after pre-testing education/counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 94 | 91 | 92 | 93
score on a scale | 16 [14 to 18] | 17 [15 to 19] | 17 [15 to 18] | 16 [15 to 18]

2. Primary Outcome: Genetic Counseling Satisfaction (Post-Test)
Description: Genetic Counseling Satisfaction Scale (GCSS) (6-item scale, score range 6-30, higher scores mean greater satisfaction)
Time Frame: Immediately after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 76 | 74 | 70 | 67
score on a scale | 24 [18 to 26.75] | 25 [20.5 to 27] | 25 [21.75 to 28] | 26 [21 to 28]

3. Primary Outcome: Test-Related Distress
Description: Revised Impact of Events Scale (22-item, score range 0-88, higher scores mean greater event-related distress)
Time Frame: 3 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 72 | 69 | 73 | 68
score on a scale | 0 [0 to 4.75] | 1 [0 to 9] | 0 [0 to 6] | 0 [0 to 5]

4. Secondary Outcome: Genetic Counseling Satisfaction (Pre-Test)
Description: Genetic Counseling Satisfaction Scale (GCSS) (6-item scale, score range 6-30, higher scores mean greater satisfaction)
Time Frame: Immediately after pre-test education/counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 93 | 90 | 89 | 88
score on a scale | 22 [20 to 26] | 23 [21 to 25.8] | 24 [21 to 27] | 25 [22 to 27.2]

5. Secondary Outcome: Depression
Description: Geriatric Depression Scale (GDS, 15-item score range 0-15, higher means greater depression)
Time Frame: 3 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 68 | 67 | 72 | 64
score on a scale | 3 [1 to 5] | 3 [1 to 4] | 2.5 [1 to 6] | 3 [2 to 5]

6. Secondary Outcome: Depression
Description: Geriatric Depression Scale (GDS, 15-item score range 0-15, higher means greater depression)
Time Frame: 6 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 62 | 65 | 70 | 61
score on a scale | 3 [1 to 5.250] | 3 [1 to 4] | 3 [1 to 6] | 3 [1 to 6]

7. Secondary Outcome: State-Trait Anxiety Index-State Score
Description: State-Trait Anxiety Index -State Score (STAI-S, 20-item, min score 20/max score 80, higher means greater anxiety). 20 of the total 40 items included in the State Score are predefined according to the validated scale.
Time Frame: 3 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 68 | 67 | 72 | 62
score on a scale | 35 [24.25 to 44.75] | 36 [25 to 41] | 35 [28 to 47.75] | 36 [26 to 44.25]

8. Secondary Outcome: State-Trait Anxiety Index -State Score
Description: State-Trait Anxiety Index -State Score (STAI-S, 20-item, min score 20/max score 80, higher means greater anxiety). 20 items of the full STAI scale that includes 40 items are predefined according to the validated scale.
Time Frame: 6 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 61 | 63 | 66 | 59
score on a scale | 35 [27 to 42.5] | 36 [29 to 44] | 34.5 [27.5 to 49] | 36 [23 to 45]

9. Secondary Outcome: State-Trait Anxiety Index -Trait Score
Description: State-Trait Anxiety Index -Trait Score (STAI-T, 20-item, min score 20/max score 80, higher means greater anxiety). 20 items of the full STAI scale that includes 40 items are predefined according to the validated scale.
Time Frame: 3 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 68 | 67 | 72 | 62
score on a scale | 34 [26 to 44] | 33 [28 to 41] | 38 [26 to 47] | 34 [27 to 42.25]

10. Secondary Outcome: State-Trait Anxiety Index -Trait Score
Description: as for outcome 9
Time Frame: 6 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 61 | 63 | 66 | 59
score on a scale | 34 [26 to 42] | 34 [27 to 43] | 35 [24 to 45] | 35 [26 to 43]

11. Secondary Outcome: Quality of Life in Parkinson's Disease
Description: Parkinsons disease quality of life scale- 39 (PDQ39). The PDQ-39 is a disease-specific health status measure that assess multiple dimensions of daily living. It is a validated, self-report measure for people with PD. Score range is from 0-100, with higher scores indicating a worse quality of life.
Time Frame: 3 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 68 | 67 | 72 | 61
score on a scale | 21.41 [10.74 to 36.76] | 15.83 [9.948 to 25.26] | 16.56 [6.315 to 32.83] | 18.44 [11.74 to 28.28]

12. Secondary Outcome: Quality of Life in Parkinson's Disease
Description: as for outcome 11
Time Frame: 6 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 61 | 63 | 66 | 59
score on a scale | 20.99 [11.35 to 34.19] | 15.31 [7.344 to 28.7] | 17.79 [7.5 to 33.82] | 19.22 [11.09 to 34.69]

13. Secondary Outcome: Test-Related Distress
Description: Revised Impact of Events Scale (22-item, score range 0-88, higher scores mean greater event-related distress)
Time Frame: 6 months after disclosure counseling
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
Number analyzed (Participants) | 68 | 67 | 73 | 67
score on a scale | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 6] | 0 [0 to 5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected at each study visit up to 6 months post disclosure, coinciding with the final study visit.
Description: AEs reviewed during the study include death during the study period or medical event during a study visit. Study outcomes were evaluated to determine AEs including number of unique individuals (not unique events) above cutpoint for psychiatric outcomes during any study visit (IES-R: above 33 point cutpoint; GDS: Above 5 point cutpoint; STAI: Above 40 on either sub scale).
Groups:
- IMAGINE-PD/Virtual: Pre-test genetic counseling through the Interactive Multimedia Approach to Genetic counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) website. Genetic results disclosure via virtual visit with a genetic counselor.
  IMAGINE-PD: The Interactive, Multimedia Approach to Genetic Counseling to INform and Educate in Parkinson's Disease (IMAGINE-PD) is a novel, interactive, web-based, audiovisual, self-guided, genetic counseling tool in the development phase. Essential genetic counseling themes, outlined by a senior certified clinical genetics counselor in accordance with national guidelines, are presented in a web-based format, utilizing videos, text, pictures, and audio. Participants can interact with IMAGINE-PD at their own pace, with the ability to move backward and forward, repeat sections, and have the ability to submit questions to the genetic counselor via e-mail.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans) within the PennChart/EPIC electronic medical record dashboard.
- Virtual/Virtual: Pre-test genetic counseling and genetic results disclosure via virtual visit with a genetic counselor.
  Virtual genetic counseling: The virtual visits will be conducted by a certified genetic counselor to provide all counseling in accordance with guidelines set forth by the National Society of Genetic Counselors. The counseling visit will be conducted in real-time on an established and secure audiovisual conferencing telemedicine platform (BlueJeans) within the PennChart/EPIC electronic medical record dashboard.
Arm/Group | IMAGINE-PD/Virtual | IMAGINE-PD/Telephone | Virtual/Telephone | Virtual/Virtual
All-Cause Mortality (participants affected / at risk) | 0/94 | 1/91 | 1/92 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/91 | 0/92 | 0/93
Other Adverse Events (participants affected / at risk) | 83/94 | 82/91 | 78/92 | 83/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMAGINE-PD/Virtual (N=94) | IMAGINE-PD/Telephone (N=91) | Virtual/Telephone (N=92) | Virtual/Virtual (N=93)
Impact of Events IES-R (Psychiatric disorders) | 5 | 7 | 2 | 6 — Unique individuals (not unique events) above outpoint for psychiatric outcomes during any study visit (IES-R: above 33 point cutpoint).
Depression (Psychiatric disorders) | 33 | 26 | 29 | 27 — Unique individuals (not unique events) above outpoint for psychiatric outcomes during any study visit (GDS: Above 5 point cutpoint)
Anxiety (Psychiatric disorders) | 45 | 49 | 46 | 50 — Unique individuals (not unique events) above outpoint for psychiatric outcomes during any study visit (STAI: Above 40 on either sub scale)
Medical event unrelated to study (General disorders) | 0 | 0 | 1 | 0 — Medical event during study visit that was unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04527146/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04527146/ICF_001.pdf